CLINICAL TRIAL: NCT05646446
Title: Integrated Alcohol and Sexual Assault Prevention for Bisexual Women
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding Terminated
Sponsor: Lifespan (Other)
Responsible Party: Principal Investigator, Lindsay Orchowski Ph.D., Associate Professor (Research), Lifespan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R34AA030035 (NIH)
Record Dates: First submitted 2022-12-05; First posted 2022-12-12 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Alcohol Use, Unspecified; Sexual Assault
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REACH Program (Experimental): The REACH program addresses alcohol use, sexual assault risk, and experiences relating to experiences of harm among bisexual women.
  Interventions: Behavioral: REACH Program
- Wait List Control Group (No Intervention): The Wait List Control Group will have the opportunity to complete the REACH program after completing study assessments at the 4-month follow-up.

INTERVENTIONS:
Behavioral: REACH Program — The REACH program addresses alcohol use, sexual assault risk, and experiences relating to harm among bisexual women.
  Arms: REACH Program

SUMMARY:
The goal of this clinical trial is to develop and evaluate the preliminary efficacy of an intervention to address reducing alcohol use, sexual revictimization, and psychological distress among bisexual+ women (i.e., attraction to more than one gender: bisexual, pansexual, queer). The main questions the study seeks to answer are: 1) what is the feasibility of the recruitment method, research design, interventionist training methods, and delivery of the intervention; 2) does the intervention, relative to control, at the 2- and 4-month follow-up period, produce reductions in the quantity and frequency of alcohol use, sexual victimization, and psychological distress (anxiety, depression). Follow-up assessments are completed at 2- and 4-months following program completion. The intervention is compared to a wait list control group.

ELIGIBILITY:
Inclusion Criteria:

* be between the ages of 18 and 24 years of age;
* identify as female gender or fluid, or gender non-conforming, gender queer, or non-binary
* identify as bisexual+ (i.e., attraction to more than one gender: bisexual, pansexual, queer);
* report a history of attempted or completed penetrative acts of sexual victimization (i.e., oral, vaginal, anal) since age 14 via coercion, incapacitation or force;
* report exceeding the national recommended limits for daily drinking (4 or more for women) on two or more occasions in the past month;
* report past month sexual activity.

Exclusion Criteria:

* current suicide risk on the Beck Depression Inventory
* current symptoms of alcohol use withdrawal on the Alcohol Use Withdrawal Checklist

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female gender or fluid, gender non-conforming, gender queer, or non-binary
Enrollment: 0 (Actual)
Dates: Start 2023-08-03 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Alcohol Use | Change from baseline alcohol use at 4 months.
  The number of past month drinking days (Minimum = 0, Maximum = 31), average drinks per drinking day (Minimum = 0, Maximum = unspecified), number of heavy drinking days (Minimum = 0, Maximum = 30), assessed via the Time Line Follow Back, with greater scores meaning worse outcomes)
Sexual Victimization | Reductions in comparison to control at 4 months.
  Assessed via the Sexual Experiences Survey. Summary score calculated that reflects both frequency and severity (Minimum = 0, Maximum = 63). Higher scores mean worse outcomes.

SECONDARY OUTCOMES:
Anxiety | Change from baseline at 4-months.
  Assessed via the Generalized Anxiety Disorder 7 (GAD-7) (Minimum = 0, Maximum = 21), with higher scores meaning worse outcomes.
Depression | Change from baseline at 4-months.
  Assessed via the Patient Health Questionnaire 9 (PHQ-9) (Minimum = 0, Maximum = 27), with higher scores meaning worse outcomes.
Mindfulness | Change from baseline at 4-months.
  Assessed via the Mindful Attention and Awareness Scale (Minimum = 15, Maximum = 90), with higher scores meaning better outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Per sponsor requirements, data will be shared using the National Institutes of Mental Health Data Archive.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The research team will submit data on or before the Data Archive submission due dates (April 1 and October 1 each year) in accordance with the applicable Data Sharing Terms and Conditions of the award.